CLINICAL TRIAL: NCT01575782
Title: Chloroquine as an Anti-autophagic Radiosensitizing Drug in Stage I-III Small Cell Lung Cancer (SCLC) Patients: a Phase I Trial.
Brief Title: Chloroquine as an Anti-autophagic Radiosensitizing Drug in Stage I-III Small Cell Lung Cancer
Acronym: Chloroquine
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Maastricht Radiation Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHLOROQUINE I-III
Record Dates: First submitted 2012-04-03; First posted 2012-04-11 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Small Cell Lung Cancer
Keywords: small cell lung cancer; stage I-III; chloroquine; Phase I
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Chloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chloroquine (Experimental)
  Interventions: Drug: Chloroquine

INTERVENTIONS:
Drug: Chloroquine — Daily intake of Chloroquine during radiotherapy
  Other Names: A-CQ 100mg per tablet

SUMMARY:
Chloroquine can make tumor cells less resistant to chemo/radiotherapy. In this trial chloroquine is given during radiotherapy. The dose is increased in cohorts of at least 3 patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed stage I-III small cell lung cancer, excluding malignant pleural/pericardial effusion.
* At least one measurable disease site, defined as lesion of ≥ 1 cm unidimensionally on CT-scan
* WHO performance status 0-2
* Absolute neutrophil count at least 1800/µl and platelets at least 100000/µl and hemoglobin at least 6.2 mmol/l.
* Adequate renal function: calculated creatinine clearance at least 60 ml/min
* Adequate hepatic function: Total bilirubin ≤ 1.5 x upper limit of normal (ULN) for the institution; ALT, AST, and alkaline phosphatase ≤ 2.5 x ULN for the institution (in case of liver metastases ≤ 5 x ULN for the institution)
* No previous platinum chemotherapy or topo-isomerase-inhibitors for SCLC.
* Lung function: FEV1 at least 30 % and DLCO at least 30 % of the age predicted value
* No history of prior chest radiotherapy
* Life expectancy more than 6 months
* Willing and able to comply with the study prescriptions
* 18 years or older
* Not pregnant or breast feeding and willing to take adequate contraceptive measures during the study
* Ability to give and having given written informed consent before patient registration
* No mixed pathology, e.g. non-small cell plus small cell cancer
* No recent (< 3 months) severe cardiac disease (NYHA class >1) (congestive heart failure, infarction)
* No history of cardiac arrythmia (multifocal premature ventricular contractions, uncontrolled atrial fibrillation, bigeminy, trigeminy, ventricular tachycardia) which is symptomatic and requiring treatment (CTC AE 3.0), or asymptomatic sustained ventricular tachycardia. Asymptomatic atrial fibrillation controlled on medication is allowed.
* No cardiac conduction disturbances or medication potentially causing them:
* QTc interval prolongation with other medications that required discontinuation of the treatment
* Congenital long QT-syndrome or unexplained sudden death of first degree relative under 40 years of age
* QT interval > 480 msec (note: when this is the case on screening ECG, the ECG may be repeated twice. If the average QT-interval of these 3 measurements remains below 480 msec, patient is eligible)
* Patients on medication potentially prolongating the QT-interval are excluded if the QT-interval is > 460 msec (Appendix, table 2).
* Medication that might cause QT-prolongation or Torsades de pointes tachycardia is not allowed (Appendix, Table 1). Drugs with a risk of prolongating the QT-interval that cannot be discontinued are allowed, however, under close monitoring by the treating physician (Appendix, table 2).
* Complete left bundle branch block
* No uncontrolled infectious disease
* No other active malignancy
* No major surgery (excluding diagnostic procedures like e.g. mediastinoscopy) in previous 4 weeks
* No treatment with investigational drugs in 4 weeks prior to or during this study
* No chronic systemic immune therapy
* No known G6PD deficiency
* Patients must not have psoriasis or porphyria.
* No known hypersensitivity to 4-aminoquinoline compound.
* Patients must not have retinal or visual field changes from prior 4-aminoquinoline compound use.
* No known prior hypersensitivity to cisplatin, etoposide or chloroquine or any of their components.

Exclusion Criteria:

- The opposite of the above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 3 months after inclusion

SECONDARY OUTCOMES:
Response of the tumour (regression, progression, stable disease) | 2 years after inclusion
Overall survival | 2 years after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Lambin, MD, PhD, Principal Investigator — Maastro Clinic, The Netherlands
Locations (1):
- MAASTRO clinic, Maastricht, Limburg, Netherlands